CLINICAL TRIAL: NCT06392633
Title: SURGERY VS BOTULINUM TOXIN ON QUALITY OF LIFE IN STROKE PATIENTS
Brief Title: SURGERY VS BOTULINUM TOXIN ON QUALITY OF LIFE IN STROKE PATIENTS: RANDOMIZED TRIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Responsible Party: Principal Investigator, Pedro Hernández Cortés, MD PhD, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI20/01574
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: spastic hand; botulinum toxin; surgery; quality of life
MeSH Terms: conditions — Stroke | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Patients who meet the inclusion criteria and who will be treated with botulinum toxin (1 injection/4months).
  Interventions: Drug: Botulinum Toxin A
- Group II (Experimental): Patients who meet the inclusion criteria and who will be treated by surgery.
  Interventions: Procedure: spastic hand sugery

INTERVENTIONS:
Procedure: spastic hand sugery — Deformity correction can be performed with single event multilevel surgery, using a combination of soft tissue releases and lengthening, tendon transfers and joint stabilization procedures. In addition, selective and supraselective neurectomies can also be performed.
  Arms: Group II
Drug: Botulinum Toxin A — Treatment consists of periodic injections of the toxin into the spastic muscles. It causes reversible chemical denervation by preventing the release of acetylcholine vesicles at the neuromuscular junctions of the affected muscles.
  Arms: Group I

SUMMARY:
We present a research project in the form of a controlled clinical trial with the aim of analyzing and demonstrating whether the surgical treatment of upper limb spasticity is an effective and efficient measure to improve dependence and quality of life perceived by patients with sequelae of stroke and therefore, should be included in the therapeutic protocols, in which it is not usually contemplated, as a complement or alternative to traditional treatment with botulinum toxin, rehabilitation and occupational therapy.

DETAILED DESCRIPTION:
Cerebrovascular accident (CVA) or "stroke" is the leading cause of permanent disability in adulthood and many patients require lifelong medical treatment and assistance from other people for the development of their daily activities. The repercussion in the family, professional, labor and social fields is enormous, producing a very important economic expense. The usual treatment of spastic upper limb secondary to stroke is rehabilitation, occupational therapy and periodic injection of botulinum toxin, and surgical correction is not usually considered. A two-arm Randomized Clinical Trial [surgical treatment (n=22) vs. botulinum toxin (n=22)] is proposed with the aim of investigating the efficacy and efficiency of surgery for upper limb spasticity with respect to treatment with botulinum toxin in patients with established spastic sequelae after stroke.

We will evaluate the effect on functionality and "hygienic" changes; the impact on quality of life, sleep quality, anxiety and depression; as well as on brain activity by Functional Magnetic Resonance Imaging, at baseline and at 6 and 12 months follow-up. The health and care costs of the established groups of patients will also be evaluated. This research is framed in the context of chronic diseases, aging and patients with functional and mobility difficulties. The results of this work are expected to have a great impact due to the high prevalence of the disease, the severe disability it causes, and the number of patients who would benefit, in addition to the savings in healthcare resources. The incorporation of surgery into stroke care would change the current treatment paradigm, favoring the formation of multidisciplinary teams for the treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age, with spasticity in the upper limb due to stroke, with a minimum evolution time of 12 months, who, after being informed orally and in writing of the objectives of the study, sign the informed consent form (themselves or their legal representatives).

Exclusion Criteria:

* Absence of consent, refusal of possible surgical treatment, stroke evolution time of less than 12 months, anaesthetic risk (ASA) class IV or higher, presence of involuntary movements, inability to respond adequately to surveys, deformities that cannot be addressed by surgical treatment or inability to follow up for at least one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life by 36-Item Short Form Survey Instrument (SF-36) | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and have been widely used.
Quality of life by Newcastle Stroke-Specific Quality of Life Measure | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  is a specific questionnaire to measure the QoL of patients who suffered a stroke. It was developed and validated by Buck et al. It is different from other questionnaires because it includes domains of vision, cognition and communication, and it can used for patients with ischaemic or haemorrhagic stroke and motor aphasia.

SECONDARY OUTCOMES:
Functional outcome by Asworth scale | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  It measures the degree of spasticity from 0 to 5. Significant improvement of at least 1 of the 5 joints evaluated (elbow, forearm, wrist, thumb, fingers) will be considered a positive result.
Functional outcome by House hand function scale | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  Scale of hand function with 10 degrees of capability
Functional outcome by Fugl-mayer scale | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  is the first quantitative evaluative instrument for measuring sensorimotor stroke recovery, based on Twitchell and Brunnstrom's concept of sequential stages of motor return in the hemiplegic stroke patient.
Functional outcome by GAS score | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  5-grade scale for the domains hygiene, esthetics and pain. Krasny-Pacini y cols, 2013
Carer Burden by Carer Burden Score | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  Scores the caregiver's degree of difficulty for 4 basic activities (nail clipping, palm grooming, armpit grooming, arm dressing) on a 5-point Likert scale.
Pain by Visual Analogue Scale | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  A tool used to help a person assess the intensity of certain sensations and feelings, such as pain. The visual analogue pain scale is a straight line where one end means no pain and the other end means the worst pain imaginable. The patient marks a point on the line that matches the amount of pain he or she feels.
Sleep health by SATED scale | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  5 questions scale about satisfaction, alertness, timing, efficiency and duration of sleep to know the sleep health of patients. Higher scores (0-10) mean better sleep health.
Anxiety and depression by HADS scale | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  Includes 14 items, with scores from 0 to 3 (higher scores reflect greater severity of symptomatology).
Activity, structure and brain function by MRI | t0 (basal assesment) t1 (6 months evaluation) t2 (12 months evaluation)
  Functional Magnetic Resonance Imaging (fMRI) at rest and with the patient's repeated attempt to extend the elbow and wrist. Anatomical and functional volumes shall be obtained by MRI and fMRI imaging, using a Siemens Prisma 3T functional MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

REFERENCES:
- [Derived] Hurtado-Olmo P, Gonzalez-Santos A, Iruela LDO, Castro-Ropero B, Zuniga-Gomez L, Bueno-Garcia AI, Guijosa-Campos P, Gomez-Pozo B, Hita-Contreras F, Hernandez-Cortes P. Impact of surgery on rehabilitation care and quality of life perceived by patient with post-stroke upper limb spasticity: Study protocol for a randomized controlled trial. PLoS One. 2025 Apr 30;20(4):e0322588. doi: 10.1371/journal.pone.0322588. eCollection 2025. PMID 40305524